CLINICAL TRIAL: NCT01965158
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Naldemedine in the Treatment of Opioid-induced Constipation in Subjects With Non-malignant Chronic Pain Receiving Opioid Therapy
Brief Title: Efficacy and Safety of Naldemedine in the Treatment of Opioid-induced Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1314V9231; 2013-002241-11 (EudraCT Number)
Record Dates: First submitted 2013-09-30; First posted 2013-10-18 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2016-04

CONDITIONS: Opioid-induced Constipation
Keywords: Opioid-induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naldemedine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naldemedine (Experimental): Participants received 0.2 mg naldemedine orally once daily for 12 weeks.
  Interventions: Drug: Naldemedine
- Placebo (Placebo Comparator): Participants received matching placebo orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naldemedine — Naldemedine 0.2 mg tablet taken orally once a day
  Other Names: S 297995; Symproic®
  Arms: Naldemedine
Drug: Placebo — Placebo tablet taken orally once a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of naldemedine in the treatment of opioid-induced constipation (OIC) in adults with non-malignant chronic pain who are not using laxatives.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 80 years inclusive at the time of informed consent
2. Subjects must have non-malignant chronic pain treated with opioids and must have opioid-induced constipation (OIC)
3. Subjects must be treated with a stable opioid regimen at a total daily dose on average of ≥ 30 mg equivalents of oral morphine sulfate
4. Subjects must not be currently using laxatives or must be willing to discontinue laxative use at Screening and must be willing to use only the rescue laxatives provided throughout the study duration
5. Subjects must meet opioid-induced constipation criteria based on the Bowel Movement and Constipation Assessment (BMCA) Diary

Exclusion Criteria:

1. Evidence of significant structural abnormalities of the gastrointestinal (GI) tract
2. Evidence of active medical diseases affecting bowel transit
3. History or presence of pelvic disorders that may be a cause of constipation
4. Surgery (except for minor procedures) within 60 days of Screening
5. History of chronic constipation prior to starting analgesic medication or any potential non-opioid cause of bowel dysfunction that may be a major contributor to the constipation (e.g., mechanical GI obstruction)
6. Subjects who have never taken laxatives for the treatment of OIC
7. History of active treatment for cancer within the last 2 years (except for basal cell or squamous cell carcinoma of the skin that have been successfully resected) or tamoxifen [Nolvadex®] and raloxifene [Evista®] when being used for prevention of breast cancer
8. Current use of any prohibited medication including opioid antagonists, partial agonists or mixed agonists/antagonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (65):
- United States (37):
  - Shionogi Research Site, Birmingham, Alabama
  - Shionogi Research Site, Phoenix, Arizona
  - Shionogi Research Site, Fresno, California
  - Shionogi Research Site, Long Beach, California
  - Shionogi Research Site, National City, California
  - Shionogi Research Site, North Hollywood, California
  - Shionogi Research Site, Oceanside, California
  - Shionogi Research Site, Golden, Colorado
  - Shionogi Research Site, Miami, Florida
  - Shionogi Research Site, Miami Springs, Florida
  - Shionogi Research Site, Orlando, Florida
  - Shionogi Research Site, Sarasota, Florida
  - Shionogi Research Site, West Palm Beach, Florida
  - Shionogi Research Site, Winter Park, Florida
  - Shionogi Research Site, Marietta, Georgia
  - Shionogi Research Site, Shreveport, Louisiana
  - Shionogi Research Site, Caro, Michigan
  - Shionogi Research Site, Flint, Michigan
  - Shionogi Research Site, Hazelwood, Missouri
  - Shionogi Research Site, Las Vegas, Nevada
  - Shionogi Research Site, Belvidere, New Jersey
  - Shionogi Research Site, East Brunswick, New Jersey
  - Shionogi Research Site, Albuquerque, New Mexico
  - Shionogi Research Site, Great Neck, New York
  - Shionogi Research Site, Hollis, New York
  - Shionogi Research Site, New Windsor, New York
  - Shionogi Research Site, Winston-Salem, North Carolina
  - Shionogi Research Site, Cincinnati, Ohio
  - Shionogi Research Site, Oklahoma City, Oklahoma
  - Shionogi Research Site, Medford, Oregon
  - Shionogi Research Site, West Reading, Pennsylvania
  - Shionogi Research Site, Chattanooga, Tennessee
  - Shionogi Research Site, Arlington, Texas
  - Shionogi Research Site, Austin, Texas
  - Shionogi Research Site, Dallas, Texas
  - Shionogi Research Site, Houston, Texas
  - Shionogi Research Site, San Antonio, Texas
- Austria (2):
  - Shionogi Research Site, Sankt Pölten
  - Shionogi Research Site, Vienna
- Czechia (5):
  - Shionogi Research Site, Hradec Králové
  - Shionogi Research Site, Liberec
  - Shionogi Research Site, Pardubice
  - Shionogi Research Site, Prague
  - Shionogi Research Site, Vysoké Mýto
- Germany (3):
  - Shionogi Research Site, Berlin
  - Shionogi Research Site, Eichstätt
  - Shionogi Research Site, Frankfurt am Main
- Poland (5):
  - Shionogi Research Site, Bialystok
  - Shionogi Research Site, Bydgoszcz
  - Shionogi Research Site, Czeladź
  - Shionogi Research Site, Gorzów Wielkopolski
  - Shionogi Research Site, Warsaw
- Spain (3):
  - Shionogi Research Site, Alicante
  - Shionogi Research Site, Cadiz
  - Shionogi Research Site, Madrid
- United Kingdom (10):
  - Shionogi Research Site, Belfast
  - Shionogi Research Site, Bexhill-on-Sea East Sussex
  - Shionogi Research Site, Crownhill Plymouth
  - Shionogi Research Site, Fowey Cornwall
  - Shionogi Research Site, Liskeard Cornwall
  - Shionogi Research Site, London
  - Shionogi Research Site, Penzance Cornwall
  - Shionogi Research Site, Saint Austell Cornwall
  - Shionogi Research Site, Soham Ely Cambs
  - Shionogi Research Site, Tomairt

REFERENCES:
- [Derived] Hale ME, Wild JE, Yamada T, Yokota T, Tack J, Andresen V, Drewes AM. Naldemedine is effective in the treatment of opioid-induced constipation in patients with chronic non-cancer pain who had a poor response to laxatives. Therap Adv Gastroenterol. 2021 Jul 31;14:17562848211032320. doi: 10.1177/17562848211032320. eCollection 2021. PMID 34377150
- [Derived] Camilleri M, Hale M, Morlion B, Tack J, Webster L, Wild J. Naldemedine Improves Patient-Reported Outcomes of Opioid-Induced Constipation in Patients with Chronic Non-Cancer Pain in the COMPOSE Phase 3 Studies. J Pain Res. 2021 Jul 16;14:2179-2189. doi: 10.2147/JPR.S282738. eCollection 2021. PMID 34295186
- [Derived] Tack J, Camilleri M, Hale M, Morlion B, Nalamachu S, Webster L, Wild J. Establishing Minimal Clinically Important Differences in Quality of Life Measures in Opioid-Induced Constipation. Clin Gastroenterol Hepatol. 2022 Apr;20(4):855-863. doi: 10.1016/j.cgh.2021.05.004. Epub 2021 Aug 5. PMID 33965574
- [Derived] Webster LR, Hale ME, Yamada T, Wild JE. A Renal Impairment Subgroup Analysis of the Safety and Efficacy of Naldemedine for the Treatment of Opioid-Induced Constipation in Patients with Chronic Non-Cancer Pain Receiving Opioid Therapy. J Pain Res. 2020 Mar 24;13:605-612. doi: 10.2147/JPR.S237833. eCollection 2020. PMID 32280263
- [Derived] Wild J, Webster L, Yamada T, Hale M. Safety and Efficacy of Naldemedine for the Treatment of Opioid-Induced Constipation in Patients with Chronic Non-Cancer Pain Receiving Opioid Therapy: A Subgroup Analysis of Patients >/= 65 Years of Age. Drugs Aging. 2020 Apr;37(4):271-279. doi: 10.1007/s40266-020-00753-2. PMID 32086791
- [Derived] Wild J, Yamada T, Arjona Ferreira JC, Hale M. Onset of action of naldemedine in the treatment of opioid-induced constipation in patients with chronic noncancer pain: results from 2 randomized, placebo-controlled, phase 3 trials. Pain. 2019 Oct;160(10):2358-2364. doi: 10.1097/j.pain.0000000000001629. PMID 31145214
- [Derived] Hale M, Wild J, Reddy J, Yamada T, Arjona Ferreira JC. Naldemedine versus placebo for opioid-induced constipation (COMPOSE-1 and COMPOSE-2): two multicentre, phase 3, double-blind, randomised, parallel-group trials. Lancet Gastroenterol Hepatol. 2017 Aug;2(8):555-564. doi: 10.1016/S2468-1253(17)30105-X. Epub 2017 May 30. PMID 28576452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 68 sites in North America and Europe, including Austria, Czech Republic, Germany, Poland, Spain, United Kingdom, and the United States.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to 0.2 mg of naldemedine or placebo. Participants were stratified based on their documented opioid use (average total daily dose (TDD) during the 14-consecutive-day qualifying period) as follows:
  * 30 to 100 mg equivalents of oral morphine sulfate
  * > 100 mg equivalents of oral morphine sulfate
Groups:
- Placebo: Participants received placebo orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Naldemedine | Placebo
Started | 274 (Includes 1 participant enrolled at 2 different sites simultaneously) | 273 (Includes 1 participant enrolled at 2 different sites simultaneously)
Received Treatment | 272 | 273
Completed | 233 | 238
Not Completed | 41 | 35
Not completed — Adverse Event | 14 | 5
Not completed — Withdrawal by Subject | 16 | 24
Not completed — Lost to Follow-up | 7 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Other - Miscellaneous | 3 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population included all randomized participants; one participant was excluded from each arm due to enrollment at 2 different sites simultaneously.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naldemedine | Placebo | Total
Number analyzed (Participants) | 273 | 272 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.44) | 53.4 (11.03) | 53.4 (10.73)
Age, Customized [Number; unit: participants]
  < 40 years | 25 | 26 | 51
  ≥ 40 to < 65 years | 209 | 199 | 408
  ≥ 65 years | 39 | 47 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 168 | 329
  Male | 112 | 104 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 247 | 245 | 492
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Black or African American | 53 | 48 | 101
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  White | 216 | 220 | 436
Stratification by Opioid Dose [Number; unit: participants] — Dose of opioid was calculated using maintenance and breakthrough morphine equivalent dose. If any participants were treated with < 30 mg, the participants were counted in '30-100 mg'.
  participants
    30-100 mg | 155 | 153 | 308
    > 100 mg | 118 | 119 | 237
Spontaneous Bowel Movements per Week [Mean (Standard Deviation); unit: spontaneous bowel movements] | 1.31 (0.746) | 1.30 (0.713) | 1.31 (0.729)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Spontaneous Bowel Movement (SBM) Response
Description: A bowel movement and constipation assessment (BMCA) was completed by participants every day during the screening and treatment periods to record information about bowel movements (BMs) and constipation. An SBM was defined as a bowel movement that occurred without the use of rescue laxative therapy during the 24 hours prior to the BM.
  A responder was defined as a participant having 9 or more positive response weeks out of the 12-week Treatment Period and 3 positive response weeks out of last 4 weeks of the 12-week Treatment Period. A positive response week was defined as ≥ 3 SBMs per week and an increase from baseline of ≥ 1 SBM per week for that week. If a participant had less than 4 days of diary entries for a week, that week was treated as a "non-response" week.
  Any participant with insufficient primary endpoint data (data for less than 9 out of 12 weeks of the Treatment Period or less than 3 out of the last 4 weeks of the 12-week Treatment Period) was treated as a non-responder.
Time Frame: 12-week treatment period
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 273 | 272
percentage of participants | 47.6 [41.6 to 53.7] | 34.6 [28.9 to 40.5]
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel — To control the overall type I error rate to be ≤ 0.05 for the primary and secondary efficacy endpoints, a fixed-sequence (hierarchical) testing approach was applied; P-value was calculated by Cochran-Mantel-Haenszel test adjusted by the opioid dose strata; Difference = 13.0, 95% CI 2-sided [4.8 to 21.3], Standard Error of Mean 4.19

2. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in the Number of Spontaneous Bowel Movements Per Week
Description: A bowel movement and constipation assessment (BMCA) was completed by participants every day during the screening and treatment periods to record information about bowel movements (BMs) and constipation. An SBM was defined as a bowel movement that occurred without the use of a rescue laxative therapy during the 24 hours prior to the BM.
  Baseline was defined as the 14 days in the screening period prior to study drug administration.
Time Frame: Baseline and the last 2 weeks of the treatment period (Weeks 11 and 12 for participants who completed 12 weeks of treatment)
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: spontaneous bowel movements / week
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 273 | 272
spontaneous bowel movements / week | 3.42 (0.193) | 2.12 (0.192)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA model has the terms for treatment group as a fixed effect and the opioid dose strata as a covariate; LS Mean Difference = 1.30, 95% CI 2-sided [0.77 to 1.83], Standard Error of Mean 0.271

3. Secondary Outcome: Change From Baseline to Week 1 in the Number of Spontaneous Bowel Movements Per Week
Description: as for outcome 2
Time Frame: Baseline and Week 1
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: spontaneous bowel movements / week
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 273 | 272
spontaneous bowel movements / week | 3.48 (0.185) | 1.36 (0.184)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA model has the terms for treatment group as a fixed effect and the opioid dose strata as a covariate; LS Mean Difference = 2.11, 95% CI 2-sided [1.60 to 2.63], Standard Error of Mean 0.260

4. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in the Number of Complete Spontaneous Bowel Movements Per Week
Description: A bowel movement and constipation assessment (BMCA) was completed by participants every day during the screening and treatment periods to record information about bowel movements (BMs) and constipation. A complete spontaneous bowel movement (CSBM) was defined as an SBM which was accompanied by the feeling of complete evacuation.
Time Frame: as for outcome 2
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: complete spontaneous BMs / week
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 273 | 272
complete spontaneous BMs / week | 2.58 (0.170) | 1.57 (0.170)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model has the terms for treatment group as a fixed effect and the opioid dose strata as a covariate; LS Mean Difference = 1.01, 95% CI 2-sided [0.54 to 1.48], Standard Error of Mean 0.240

5. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in the Number of Spontaneous Bowel Movements With No Straining Per Week
Description: A bowel movement and constipation assessment (BMCA) was completed by participants every day during the screening and treatment periods to record information about bowel movements (BMs) and constipation.
  The severity of straining with each bowel movement was assessed on the following scale: 0=no straining, 1=mild straining, 2=moderate straining, 3=severe straining, 4=very severe straining. SBMs without straining were defined as SBMs with a straining score of 0.
Time Frame: as for outcome 2
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: SBMs with no straining / week
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 273 | 272
SBMs with no straining / week | 1.46 (0.141) | 0.73 (0.140)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA; The ANCOVA model has the terms for treatment group as a fixed effect and the opioid dose strata as a covariate; LS Mean Difference = 0.73, 95% CI 2-sided [0.34 to 1.12], Standard Error of Mean 0.198

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 28 days after the last dose of study drug (16 weeks).
Description: The Safety Population included all randomized participants who received at least 1 dose of study drug. One participant was excluded from each arm due to simultaneous enrollment at 2 different sites.
Arm/Group | Naldemedine | Placebo
Serious Adverse Events (participants affected / at risk) | 14/271 | 5/272
Other Adverse Events (participants affected / at risk) | 29/271 | 11/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naldemedine (N=271) | Placebo (N=272)
Appendicitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 0
Device failure (General disorders) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naldemedine (N=271) | Placebo (N=272)
Abdominal pain (Gastrointestinal disorders) | 16 | 5
Diarrhoea (Gastrointestinal disorders) | 18 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.